CLINICAL TRIAL: NCT06637033
Title: The Impact of Chewing Food on Stroke Patients With Dysphagia: A Randomized Controlled Trial
Brief Title: The Impact of Chewing Food on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babujinaya Cela (Other Government)
Responsible Party: Sponsor-Investigator, Babujinaya Cela, The Research Director, Buraidah Central Hospital
Organization: Buraidah Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jujue-stroke
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing Food Group (Experimental): This group will be given routine rehabilitation training, oral tube feeding and Chewing Food training with real food for 15 days.
  Interventions: Behavioral: Chewing Real Food; Behavioral: routine rehabilitation therapy; Behavioral: Oral tube feeding
- Control Group (Active Comparator): This group will be given routine rehabilitation training, oral tube feeding and Chewing Food training with lotus root powder for 15 days.
  Interventions: Behavioral: routine rehabilitation therapy; Behavioral: Oral tube feeding; Behavioral: Chewing Lotus Root Powder Food

INTERVENTIONS:
Behavioral: Chewing Real Food — Daily foods like candies and dumplings will be cut into small pieces. Patients will chew them before each rehabilitation training and then spit them out, with each training session lasting ten minutes.
  Arms: Chewing Food Group
Behavioral: routine rehabilitation therapy — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
Behavioral: Oral tube feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
Behavioral: Chewing Lotus Root Powder Food — Lotus Root Powder Food will be cut into small pieces. Patients will chew them before each rehabilitation training and then spit them out, with each training session lasting ten minutes.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to explore the effect of Chewing Food on quality of life and nutritional status in ischemic stroke patients. Patients will be randomly divided into an interventional group and a control group, all receiving routine rehabilitation treatment and enteral nutrition feeding. On this basis, the interventional group will receive Chewing Food training before each feeding for 10 min. Researchers will compare changes in quality of life, and nutritional status of two groups of patients before and after the study to see if Chewing Food can improve the quality of life and nutritional status in ischemic stroke patients.

DETAILED DESCRIPTION:
The study will last 15 days for each participant. The goal of this clinical trial is to explore the effect of Chewing Food on quality of life and nutritional status in ischemic stroke patients. Patients will be randomly divided into an interventional group and a control group, all receiving routine rehabilitation treatment and enteral nutrition feeding. On this basis, the interventional group will receive Chewing Food training before each feeding for 10 min. Researchers will compare changes in quality of life, and nutritional status of two groups of patients before and after the study to see if Chewing Food can improve the quality of life and nutritional status in ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Modified Barium Swallow Impairment Profile | Day 1 and day 15
  The Modified Barium Swallow Impairment Profile is used to assess the clinical severity of oropharyngeal dysphagia. It includes 16 items and incorporates a standard Modified Barium Swallow test and is based on the gold standard of swallowing function assessment, Videofluoroscopic Swallowing Studies. The total score could range from 0 to 51, with higher scores indicating more severe oropharyngeal dysphagia.

SECONDARY OUTCOMES:
Dysphagia Handicap Index | Day 1 and day 15
  The Dysphagia Handicap Index is a 25-item scale to evaluate swallowing-related quality of life. The scale scores range between 0 to 100 and a higher score indicate better quality of life
Penetration-Aspiration Scale | Day 1 and day 15
  The Penetration-Aspiration Scale is used to evaluate airway protection. The level could range between 0 and 8, with higher scores indicating poor swallowing safety.
7-item Generalized Anxiety Disorder | Day 1 and day 15
  The 7-item Generalized Anxiety Disorder is used to assess anxiety. The total score could range from 0 to 21, with higher scores indicating more severe anxiety.
Stroke Self-Efficacy Questionnaire | Day 1 and day 15
  Stroke Self-Efficacy Questionnaire is used to assess self-efficacy in functional independence and self-management. The total score could range from 0 to 130. A Higher score indicated better self-efficacy.
Rehabilitation adherence | Day 1 and day 15
  Rehabilitation adherence is assessed using a 0-10 visual analog scale. The question is "How would you rate your current acceptance and compliance with rehabilitation training, where 10 is the highest and 0 is the lowest?"

CONTACTS AND LOCATIONS:
Overall Officials: Hongji Zeng, PhD, Principal Investigator — ZZU First Hospital
Locations (2):
- China (2):
  - Renmin Hospital of SND, Suzhu
  - ZZU No.1 Hospital, Zhenzhou